CLINICAL TRIAL: NCT04699981
Title: Can the Relative Fecal Abundance of BLSE and the Digestive Microbiota be Predictive of the Risk of Infection in a Carrier Patient?
Acronym: COPROBLSE2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: COPROBLSE2
Record Dates: First submitted 2020-12-30; First posted 2021-01-07 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Enterobacteria Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Patients colonized rectally with ESBL-producing enterobacteria without antibiotic pressure (Experimental): Known patients colonized rectally with ESBL-producing enterobacteria and not subjected to antibiotic pressure
  Interventions: Other: Control (Patients colonized rectally with ESBL-producing enterobacteria without antibiotic pressure)
- Case: Patients colonized rectally with ESBL-producing enterobacteriaceae, with antibiotic pressure (Experimental): Known patients colonized rectally with ESBL-producing enterobacteriaceae and subjected to antibiotic pressure (antibiotic therapy predicted greater than 24 hours) with beta-lactams or dual therapy comprising a beta-lactam. The prescription of antibiotic therapy, a decision independent of the study procedures, will be carried out as part of routine care in the context of microbiologically documented infection. The choice of molecules will be left to the discretion of clinicians.
  Interventions: Other: Case (Patients colonized rectally with ESBL-producing enterobacteriaceae, with antibiotic pressure)

INTERVENTIONS:
Other: Control (Patients colonized rectally with ESBL-producing enterobacteria without antibiotic pressure) — For patients included in the "Control group" on discharge from hospitalization and 60 days after inclusion of patients, data will be collected either from the patient's medical file (T1Control) or during '' a telephone call from the patient (T2Control). The data collected concerns the occurrence of an infectious episode. They will also benefit from a stool sample at T1 control in order to assess the evolution kinetics of the relative fecal abundance of ESBL-producing enterobacteria in these patients who are not subjected to antibiotic pressure but subjected to other drug pressures (PPI, corticosteroids, etc.).
  Arms: Control: Patients colonized rectally with ESBL-producing enterobacteria without antibiotic pressure
Other: Case (Patients colonized rectally with ESBL-producing enterobacteriaceae, with antibiotic pressure) — A stool culture is performed on the first stool emitted after the start of antibiotic therapy. 72 hours after the start of antibiotic therapy, a blood sample (5 ml) and a stool sample will be taken. A stool sample will be taken at the end of the antibiotic therapy and 60 days after the end of the antibiotic therapy. In the event of "normal" transit (daily bowel movements), the stool emitted 48 hours after the start of antibiotic therapy will be analyzed. If the patient does not pass stool, an eswab rectal swab will be taken. In the event of discharge from the hospital before the end of the antibiotic therapy and / or the D60 after the end of the antibiotic therapy, the patient will be given a prescription and an appointment at the collection center of the center concerned for the sample stool.
  Arms: Case: Patients colonized rectally with ESBL-producing enterobacteriaceae, with antibiotic pressure

SUMMARY:
Among Enterobacteriaceae, the production of beta-lactamases (ESBLs) is the leading cause of multi-resistance. The first cases of ESBL-producing Enterobacteriaceae (E-ESBL) infections were described in the 1980s and subsequently experienced worldwide dissemination.

Since the turn of the century, the prevalence of E-ESBL infections, especially among Escherichia coli (E. coli) and Klebsiella pneumoniae (K. pneumoniae) has increased dramatically.

The emergence of multidrug-resistant Enterobacteriaceae is currently a real public health problem. The European Antimicrobial Resistance Surveillance Network evaluated, among clinical strains, the rate of resistance to 3rd generation cephalosporins (C3G) at 9.5% for E. coli and 28% for K. pneumoniae. Numerous studies have shown that bacterial colonization is the prerequisite for the occurrence of many infections.

However, the existence of prior colonization does not seem to be the only risk factor for the occurrence of a secondary infection. Therefore, in patients with multidrug-resistant Gram-negative bacillus gastrointestinal carriage there appear to be factors associated with the onset of infection. Several studies have examined the risk factors associated with E-ESBL-related infections in both community-based and healthcare-associated / nosocomial infections. Two main risk factors seem to be associated with E-ESBL infections: prior antibiotic therapy and the existence of invasive devices.

A recent study, carried out on 1288 patients and aimed at validating a predictive score for the occurrence of ESBL-E bacteremia, demonstrated 5 factors associated with the appearance of E-ESBL-linked bacteremia. These factors were: (i) a history of colonization / infection with ESBL-E, (ii) age ≥ 43 years, (iii) recent hospitalization in a region with a high prevalence of ESBL-E, (iv) antibiotic therapy ≥ 6 days in the previous 6 months and (v) the existence of a chronic vascular access.

Recently, a retrospective case-control study conducted in the United States by Augustine et al. Suggested that 5% of cases of bacteremia were related to ESBL-E.

Few studies have looked at risk factors for infection in patients known to be colonized by the digestive system. In a retrospective case-control study, conducted outside the intensive care unit and including pediatric and adult patients, the authors identified 2 factors associated with the occurrence of Ec-ESBL infection in previously colonized patients. These two factors were the prior use of antibiotics with β-lactam antibiotics and β-lactamase inhibitor (s), and urinary catheterization.

In intensive care hospital patients, the occurrence of ESBL-producing enterobacteriaceae infection appears to be a rare event, including in colonized patients.

The work of Ruppé et al. showed a direct link between relative fecal abundance of EScher-producing Escherichia coli and prior antibiotic intake.

This work also demonstrated a link between the value of the relative fecal abundance in Ec-ESBL and the occurrence of a urinary tract infection linked to the same clone. In particular, the authors found that women with a low relative fecal abundance rate (≤ 0.1%) had no risk of developing an Escherichia coli urinary tract infection. Conversely, the risk increased with the relative fecal abundance of Escherichia coli, but with a positive predictive value limited to 57% for relative fecal abundances between 10 and 100%.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years old) hospitalized at the Paris Saint-Joseph Hospital Group or in the intensive care unit of Avicenne hospital, Necker Enfants Malades hospital, Center Sud Francilien, detected as a carrier of enterobacteriaceae in the digestive system ESBL producers
* Patient affiliated to a health insurance plan
* French-speaking patient
* Patient living at home, in EHPAD or retirement home
* Patient or Relative able to give free, informed and express consent

Exclusion Criteria:

* Known patient colonized rectally with ESBL-producing enterobacteria and subjected to antibiotic pressure other than beta-lactams
* Patient participating simultaneously in other intervention research that may interfere with the objectives of the study
* Patient under guardianship or curatorship
* Patient deprived of liberty
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of EBLSE | Day 60
  This outcome corresponds to comparison of the relative fecal abundance (expressed as a percentage) of ESBL E and the microbiota in the 2 groups of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit PILMIS, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (4):
- France (4):
  - Groupe Hospitalier Paris Saint-Joseph, Paris, Groupe Hospitalier Paris Saint-Joseph
  - Hôpital Necker-Enfants malades, Paris, Groupe Hospitalier Paris Saint-Joseph
  - Hôpital Avicenne, Bobigny
  - Centre Hospitalier Sud-Francilien, Corbeil-Essonnes

REFERENCES:
- [Result] Wertheim HF, Vos MC, Ott A, van Belkum A, Voss A, Kluytmans JA, van Keulen PH, Vandenbroucke-Grauls CM, Meester MH, Verbrugh HA. Risk and outcome of nosocomial Staphylococcus aureus bacteraemia in nasal carriers versus non-carriers. Lancet. 2004 Aug 21-27;364(9435):703-5. doi: 10.1016/S0140-6736(04)16897-9. PMID 15325835
- [Result] Bruyere R, Vigneron C, Bador J, Aho S, Toitot A, Quenot JP, Prin S, Charles PE. Significance of Prior Digestive Colonization With Extended-Spectrum beta-Lactamase-Producing Enterobacteriaceae in Patients With Ventilator-Associated Pneumonia. Crit Care Med. 2016 Apr;44(4):699-706. doi: 10.1097/CCM.0000000000001471. PMID 26571186
- [Result] Dubinsky-Pertzov B, Temkin E, Harbarth S, Fankhauser-Rodriguez C, Carevic B, Radovanovic I, Ris F, Kariv Y, Buchs NC, Schiffer E, Cohen Percia S, Nutman A, Fallach N, Klausner J, Carmeli Y; R-GNOSIS WP4 Study Group. Carriage of Extended-spectrum Beta-lactamase-producing Enterobacteriaceae and the Risk of Surgical Site Infection After Colorectal Surgery: A Prospective Cohort Study. Clin Infect Dis. 2019 May 2;68(10):1699-1704. doi: 10.1093/cid/ciy768. PMID 30204851
- [Result] Zahar JR, Lesprit P, Ruckly S, Eden A, Hikombo H, Bernard L, Harbarth S, Timsit JF, Brun-Buisson C; BacterCom Study Group. Predominance of healthcare-associated cases among episodes of community-onset bacteraemia due to extended-spectrum beta-lactamase-producing Enterobacteriaceae. Int J Antimicrob Agents. 2017 Jan;49(1):67-73. doi: 10.1016/j.ijantimicag.2016.09.032. Epub 2016 Nov 16. PMID 27890442
- [Result] Rodriguez-Bano J, Navarro MD, Retamar P, Picon E, Pascual A; Extended-Spectrum Beta-Lactamases-Red Espanola de Investigacion en Patologia Infecciosa/Grupo de Estudio de Infeccion Hospitalaria Group. beta-Lactam/beta-lactam inhibitor combinations for the treatment of bacteremia due to extended-spectrum beta-lactamase-producing Escherichia coli: a post hoc analysis of prospective cohorts. Clin Infect Dis. 2012 Jan 15;54(2):167-74. doi: 10.1093/cid/cir790. Epub 2011 Nov 4. PMID 22057701
- [Result] Goodman KE, Lessler J, Cosgrove SE, Harris AD, Lautenbach E, Han JH, Milstone AM, Massey CJ, Tamma PD; Antibacterial Resistance Leadership Group. A Clinical Decision Tree to Predict Whether a Bacteremic Patient Is Infected With an Extended-Spectrum beta-Lactamase-Producing Organism. Clin Infect Dis. 2016 Oct 1;63(7):896-903. doi: 10.1093/cid/ciw425. Epub 2016 Jun 28. PMID 27358356
- [Result] Augustine MR, Testerman TL, Justo JA, Bookstaver PB, Kohn J, Albrecht H, Al-Hasan MN. Clinical Risk Score for Prediction of Extended-Spectrum beta-Lactamase-Producing Enterobacteriaceae in Bloodstream Isolates. Infect Control Hosp Epidemiol. 2017 Mar;38(3):266-272. doi: 10.1017/ice.2016.292. Epub 2016 Dec 19. PMID 27989244